CLINICAL TRIAL: NCT00187993
Title: Growth Hormone Treatment of Young Adults Deficient in Growth Hormone Since Childhood : Study of Body Composition Modifications.
Brief Title: Growth Hormone Treatment of Young Growth Hormone-Deficient Adults
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Angers (Other Government)
Collaborators: Novo Nordisk A/S (Industry)
Other Study IDs: CP-04-03; 2004/10 (CCPPRB); 0673 (AFSSAPS)
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2005-09-16 (Estimated); Status verified 2005-09

CONDITIONS: Growth Hormone Deficiency
Keywords: growth hormone deficiency; growth hormone; energy expenditure; body composition
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — Growth Hormone

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

INTERVENTIONS:
Drug: Growth hormone

SUMMARY:
Hypopituitary adults with all the hormonal deficiencies are well subsituted excepted for the growth hormone (GH) and died earlier than the rest of the population. GH deficiency involves a fat mass increase with regard to lean mass, an atherogenic lipidic profile and participating to osteopenia mechanism and decrease the life quality. All these dysfunctions are partially or totally corrected by the GH prescription with patient deficient since adulthood.

However, for patients deficient since childhood, no study have demonstrated that GH treatment during childhood present these same benefit when they are treated during adulthood.

Primary objective of this study is to examine that fat mass significantly decrease due to GH treatment in adulthood for patient GH deficient since childhood, treated by GH during childhood but stopped since the end of adolescence.

We compare the body composition and others energetic metabolism parameters in two patient groups, one treated by GH during 18 months, and the other with no treatment. Body composition and bone density are measured by pletysmography (DEXA). Metabolic parameters are : energetic balance (energy intake evaluation by questionnaire, energetic expenditure evaluated by doubly labelled water) and biologic parameters (lipidic profile, thyroid hormones).

This study will evaluate if the GH treatment of young GH deficient adults since childhood can be a benefit for body composition, lipidic profile and bone density.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age > 18-35 years)
* Stable body mass +/- 5 kg in 3 months
* GH deficiency since childhood, treated by GH during childhood, having stopped GH treatment at the end of adolescence
* Want to receive again GH treatment or refusing new GH treatment
* GH deficiency confirmed at adulthood by GHRH-Arginine test
* Women receiving GH treatment must have a efficient contraceptive method
* Have given a writing informed consent

Exclusion Criteria:

* Somatotropic insufficiency
* All pathologies or treatment modifing energetic metabolism, excepted diabet mellitus and obesity
* Participating to another clinical trial during the three months befor inclusion
* Pathologies modifing bone metabolism
* Pregnancy/Feeding
* Refusal to consent

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30
Dates: Start 2005-05; Study Completion 2005-08

CONTACTS AND LOCATIONS:
Overall Officials: Rohmer Vincent, Professor, Study Director — CHU of Angers
Locations (6):
- France (6):
  - UH of Angers, Angers
  - UH of Brest, Brest
  - UH of Caen, Caen
  - UH of Limoges, Limoges
  - UH of Rennes, Rennes
  - UH of Tours, Tours